CLINICAL TRIAL: NCT02832427
Title: The First Planned Outpatient Review After Cardiac Surgery: Is Six Weeks Too Long?
Brief Title: Is Six Weeks Too Long for First Outpatient Review After Cardiac Surgery?
Acronym: FORCAST6
Status: Completed | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 203366
Record Dates: First submitted 2016-04-26; First posted 2016-07-14 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Postoperative; Dysfunction Following Cardiac Surgery
Keywords: Coronary artery bypass grafting; Heart valve surgery; Postoperative morbidity; Operative mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Although the first outpatient review following cardiac surgery is conventionally scheduled for six weeks after hospital discharge, there is no evidence to support this practice. Thirty-day mortality and morbidity rates, which are now widely used as indicators of the quality of surgical care, reveal rates that are higher than corresponding in-hospital rates. Secondly, the rates for mortality and morbidity occurring up to 6 weeks after surgery are not known. The objectives of our study are to determine the postoperative mortality and morbidity rates in the 6-week interval between hospital discharge and the first planned specialist review after cardiac surgery, and to assess the level of patient satisfaction with current practice.

The study will enrol eligible patients who are undergoing elective and urgent coronary artery bypass and/or valve surgery at our institution over a 6-month period and provide them with study information. Prior to discharge after surgery, prospective participants will be consented and given a questionnaire to take home, complete and bring along to the outpatient appointment.

The investigators will analyse the data to determine the rates and timing of the complications, and the impact on postoperative recovery. The investigators will also assess the level of patient satisfaction with the current practice.

Appropriate conclusions either in support of current practice or, a change in practice would be drawn..

DETAILED DESCRIPTION:
Rationale and Background In current practice, patients who have undergone cardiac surgery return to the outpatient clinic for their first postoperative review by the specialist team, six weeks after hospital discharge. However, there is no evidence to show that this is the optimal interval before these patients with ongoing risks of postoperative complications are reviewed. Not infrequently, after hospital discharge, cardiac surgery patients make unplanned hospital visits and/or require readmission during the 6-week wait for outpatient review due to surgery-related complications [1-3]. Whereas it is well established that 30-day mortality and morbidity rates after surgery are in excess of the corresponding in-hospital rates [4], the 42-day incidence of these postoperative complications before outpatient review, is not known. In fact the 30-day readmission and mortality rates are widely used as indicators of the quality of surgical care [5, 6], and 30-day hospital readmission rates after cardiac surgery as high as 49% has been reported [7]. It can be argued the long interval between hospital discharge and the first outpatient specialist review exposes patients to ongoing risks which explain the higher rates of surgery-related complications over time. Postoperative programmes that have incorporated cardiac surgery nurse home visits before outpatient review report significant reduction in hospital readmissions [8].

Hospital readmissions contribute significantly to healthcare costs whilst compromising the quality of care [9, 10]. As a result strategies directed at reducing 30-day adverse outcomes and readmissions have focussed on the identification of predictors of readmission and their management [11-16]. The risk factors identified older age and co-morbidities which are prevalent among patients undergoing cardiac surgery in the current era; an even stronger reason to re-examine the long-standing outpatient follow-up practice.

The purpose of this prospective observational study will be to assess the burden of postoperative mortality and morbidity in the 6-week interval between hospital discharge and the first planned outpatient review after cardiac surgery. This data will be helpful in determining if the current timing of follow-up review should be revised.

The proposed study, will seek to answer these questions and provide scientific evidence to support clinical practice.

Study goals and objectives After hospital discharge, patients who have undergone cardiac surgery still develop complications which can impair their recovery and sometimes require unplanned visits to accident and emergency departments, and hospital admissions.

The main study goal is to define the magnitude of ongoing postoperative complications suffered by discharged cardiac surgery patients before their first planned review.

Study design The study is a prospective observational study that will involve administering a questionnaire to consecutive adult patients who will undergone coronary artery bypass and/or valve surgery at our institution over a 6-month period.

Methodology On admission for surgery, eligible participants will be approached and provided with study information. Prior to discharge after surgery, prospective participants will be consented and given the study questionnaire to take home to complete themselves or by their spouse/carer.

Preoperative and peri-operative data will be collected using the standard cardiothoracic surgery electronic database programme (Patient Analysis and Tracking System), as is routine at the investigators' institution. In addition, post discharge data relating to planned and unplanned hospital attendance and/or admission, and any intervention by General Practitioner/Practice nurse during the 6 week interval before the first planned specialist review, shall be prospectively collected using the study questionnaire.

Statistical analyses The data obtained from the study questionnaire will be linked with the peri-operative data in the cardiothoracic database, managed by dedicated and specially trained staff. The database is password-protected and access to the data is restricted.

The data will be anonymised and the variables coded for statistical analyses. The analyses will include the determination of rates of different complications and the impact on the postoperative recovery. The timing of the complications/intervention will be represented on a frequency plot.

Results The study findings will be discussed at local and international scientific meetings and published in specialty journals.

The result will be used to generate hypothesis to support the application for a randomised clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing coronary artery bypass and/or valve surgery.
* Patients who can read and write in English

Exclusion Criteria:

* Postoperative stroke with neurologic deficit

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing coronary artery bypass grafting and/or valve surgery
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
The proportion of participants with postoperative mortality, or complications who require further interventions and hospital readmission . | 6 weeks
  Patients who require further interventions and hospital readmission.

SECONDARY OUTCOMES:
The timing of postoperative mortality | 6 weeks
  The postoperative mortality of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dumbor Ngaage, MS, FRCS, Principal Investigator — Castle Hill Hospital, Kingston-Upon-Hull, HU16 5JQ, UK
Locations (1):
- Castle Hill Hospital, Hull, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available.

REFERENCES:
- [Background] Shroyer AL, Coombs LP, Peterson ED, Eiken MC, DeLong ER, Chen A, Ferguson TB Jr, Grover FL, Edwards FH; Society of Thoracic Surgeons. The Society of Thoracic Surgeons: 30-day operative mortality and morbidity risk models. Ann Thorac Surg. 2003 Jun;75(6):1856-64; discussion 1864-5. doi: 10.1016/s0003-4975(03)00179-6. PMID 12822628
- [Background] Fox JP, Suter LG, Wang K, Wang Y, Krumholz HM, Ross JS. Hospital-based, acute care use among patients within 30 days of discharge after coronary artery bypass surgery. Ann Thorac Surg. 2013 Jul;96(1):96-104. doi: 10.1016/j.athoracsur.2013.03.091. Epub 2013 May 21. PMID 23702228
- [Background] Hannan EL, Zhong Y, Lahey SJ, Culliford AT, Gold JP, Smith CR, Higgins RS, Jordan D, Wechsler A. 30-day readmissions after coronary artery bypass graft surgery in New York State. JACC Cardiovasc Interv. 2011 May;4(5):569-76. doi: 10.1016/j.jcin.2011.01.010. PMID 21596331
- [Background] Siregar S, Groenwold RH, de Mol BA, Speekenbrink RG, Versteegh MI, Brandon Bravo Bruinsma GJ, Bots ML, van der Graaf Y, van Herwerden LA. Evaluation of cardiac surgery mortality rates: 30-day mortality or longer follow-up? Eur J Cardiothorac Surg. 2013 Nov;44(5):875-83. doi: 10.1093/ejcts/ezt119. Epub 2013 Mar 7. PMID 23471150
- [Background] Hwang YJ, Minnillo BJ, Kim SP, Abouassaly R. Assessment of healthcare quality metrics: Length-of-stay, 30-day readmission, and 30-day mortality for radical nephrectomy with inferior vena cava thrombectomy. Can Urol Assoc J. 2015 Mar-Apr;9(3-4):114-21. doi: 10.5489/cuaj.2547. PMID 26085868
- [Background] Shih T, Dimick JB. Reliability of readmission rates as a hospital quality measure in cardiac surgery. Ann Thorac Surg. 2014 Apr;97(4):1214-8. doi: 10.1016/j.athoracsur.2013.11.048. Epub 2014 Feb 1. PMID 24492060
- [Background] Lahey SJ, Campos CT, Jennings B, Pawlow P, Stokes T, Levitsky S. Hospital readmission after cardiac surgery. Does "fast track" cardiac surgery result in cost saving or cost shifting? Circulation. 1998 Nov 10;98(19 Suppl):II35-40. PMID 9852877
- [Background] Hall MH, Esposito RA, Pekmezaris R, Lesser M, Moravick D, Jahn L, Blenderman R, Akerman M, Nouryan CN, Hartman AR. Cardiac surgery nurse practitioner home visits prevent coronary artery bypass graft readmissions. Ann Thorac Surg. 2014 May;97(5):1488-93; discussion 1493-5. doi: 10.1016/j.athoracsur.2013.12.049. Epub 2014 Mar 6. PMID 24612701
- [Background] Lawson EH, Hall BL, Louie R, Ettner SL, Zingmond DS, Han L, Rapp M, Ko CY. Association between occurrence of a postoperative complication and readmission: implications for quality improvement and cost savings. Ann Surg. 2013 Jul;258(1):10-8. doi: 10.1097/SLA.0b013e31828e3ac3. PMID 23579579
- [Background] Wick EC, Shore AD, Hirose K, Ibrahim AM, Gearhart SL, Efron J, Weiner JP, Makary MA. Readmission rates and cost following colorectal surgery. Dis Colon Rectum. 2011 Dec;54(12):1475-9. doi: 10.1097/DCR.0b013e31822ff8f0. PMID 22067174
- [Background] Stewart RD, Campos CT, Jennings B, Lollis SS, Levitsky S, Lahey SJ. Predictors of 30-day hospital readmission after coronary artery bypass. Ann Thorac Surg. 2000 Jul;70(1):169-74. doi: 10.1016/s0003-4975(00)01386-2. PMID 10921703
- [Background] Hannan EL, Racz MJ, Walford G, Ryan TJ, Isom OW, Bennett E, Jones RH. Predictors of readmission for complications of coronary artery bypass graft surgery. JAMA. 2003 Aug 13;290(6):773-80. doi: 10.1001/jama.290.6.773. PMID 12915430
- [Background] Price JD, Romeiser JL, Gnerre JM, Shroyer AL, Rosengart TK. Risk analysis for readmission after coronary artery bypass surgery: developing a strategy to reduce readmissions. J Am Coll Surg. 2013 Mar;216(3):412-9. doi: 10.1016/j.jamcollsurg.2012.11.009. Epub 2013 Jan 11. PMID 23313544
- [Background] Billah B, Reid CM, Shardey GC, Smith JA. A preoperative risk prediction model for 30-day mortality following cardiac surgery in an Australian cohort. Eur J Cardiothorac Surg. 2010 May;37(5):1086-92. doi: 10.1016/j.ejcts.2009.11.021. Epub 2010 Feb 8. PMID 20117015
- [Background] Lancaster E, Postel M, Satou N, Shemin R, Benharash P. Introspection into institutional database allows for focused quality improvement plan in cardiac surgery: example for a new global healthcare system. Am Surg. 2013 Oct;79(10):1040-4. PMID 24160795
- [Background] Shahian DM, He X, O'Brien SM, Grover FL, Jacobs JP, Edwards FH, Welke KF, Suter LG, Drye E, Shewan CM, Han L, Peterson E. Development of a clinical registry-based 30-day readmission measure for coronary artery bypass grafting surgery. Circulation. 2014 Jul 29;130(5):399-409. doi: 10.1161/CIRCULATIONAHA.113.007541. Epub 2014 Jun 10. PMID 24916208
- See also: Publication Link — https://bjcardio.co.uk/2019/02/is-six-weeks-too-long-for-the-first-outpatient-review-after-cardiac-surgery-forcast6/